CLINICAL TRIAL: NCT04989608
Title: Cognitive Profile and Correlates in Neuroimaging After a Transient Ischemic Accident
Brief Title: Correlation Between Cognition and Neuroimaging in TIA Patients
Acronym: COG-TIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-134
Record Dates: First submitted 2021-07-22; First posted 2021-08-04 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Transient Ischemic Accident
MeSH Terms: interventions — Neuroimaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients having suffered to transient ischemic accident (Other)
  Interventions: Other: Neuroimaging
- healthy volunteers (Other)
  Interventions: Other: Neuroimaging

INTERVENTIONS:
Other: Neuroimaging — realization of a neuroimaging 1 and 3 years after the transient ischemic accident

SUMMARY:
Context:

Cognitive impairment is common after a stroke. Out of 100 patients who have suffered a stroke, 50 will develop cognitive impairment. For 16 of them, they will be responsible for an impact on autonomy (major cognitive disorder). They are conventionally attributed either to the location of the lesions or to their general volume. However, recent literature emphasizes the presence of cognitive impairment after a transient ischemic attack (TIA), when by definition the symptoms are transient and imaging without recent ischemic injury. The mechanisms of cognitive impairment in TIA are therefore poorly understood at present. There is evidence in animal models and humans for persistent brain toxicity from ischemia even in the absence of established necrosis. However, to what extent this toxicity may explain the cognitive impairment seen in TIA is not known. Indeed, the latter could just as much have the effect of vascular risk factors which significantly increase cognitive risk even in the absence of an acute event.

Objective:

The objective of the Cog-TIA program is therefore to identify whether the transient ischemic attack may be responsible for long-term structural changes in neuroimaging in the ischemic territory and whether these changes are correlated with changes in cognitive efficiency.

Material and methods:

The project is based on the Normandy-Stroke population cohort which includes patients from Caen and the surrounding area who have had a stroke or TIA. The protocol provides for neuropsychological tests evaluating the main cognitive domains at 1 year and 3 years after the initial event. The Cog-TIA project is designed as an ancillary study to the Normandy-Stroke project with the objective of including 50 patients from this cohort who presented with a transient ischemic attack. Each patient will receive a structural MRI at the same time as the neuropsychological assessments scheduled for the Normandy-Stroke study. Analyzes will be performed from T1 sequences, Proton density with centered on the hippocampus and diffusion tensors. For the T1 and proton density sequences, the analyzes will compare the volumes of the different structures longitudinally (in particular: the total hippocampal volume and of the subfields, lobar, thalamic and pallidal volumes). For the diffusion tensor analyzes, the anisotropy maps will be compared longitudinally. For each structure showing significant variation during follow-up, correlations will be made with the decline in performance on neuropsychological tests calculated using composite scores. Cognitive decline may be partly attributed to TIA if it is correlated with abnormalities in the affected hemisphere.

ELIGIBILITY:
Inclusion Criteria:

Transient ischemic accident Group

* Patient over 60 years of age with a transient ischemic attack (focal neurological deficit of less than 24 hours without ischemic injury on diffusion MRI performed in the week following the event.)
* Patient having signed a free and informed consent to participate in the Normandy-Stroke cohort.

Control group

* Subject over 60 years old
* Subject included in the Medit-AGEING research protocol
* Subject with one or more risk factor (s) for cerebrovascular disease
* Subject not opposing the use of their data for the Cog-Tia study

Non inclusion criteria

Transient ischemic accident Group

* Patient with contraindications to performing a brain MRI
* Neurological co-morbidity (history of severe head trauma, dementia, brain tumor, stroke, psychosis)
* Refusal to participate in the Normandy-Stroke cohort
* Persons deprived of their liberty by a judicial or administrative decision, persons undergoing psychiatric care, persons admitted to a health or social establishment for purposes other than that of research
* Adult persons subject to a legal protection measure or unable to express their consent

Control group

- Subject refusing to the use of their data for the Cog-Tia study

Exclusion Criteria:

* New stroke during the study participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-17 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
correlation coefficients between variations in cognitive performance assessed from a composite neuropsychological score and structural modifications | 1 year after the transient ischemic accident
  Calculation of correlation coefficients between variations in cognitive performance assessed from a composite neuropsychological score and structural modifications
correlation coefficients between variations in cognitive performance assessed from a composite neuropsychological score and structural modifications | 3 years after the transient ischemic accident
  Calculation of correlation coefficients between variations in cognitive

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France